CLINICAL TRIAL: NCT00383851
Title: A Randomized Phase II Trial of ATN-224 in Combination With Temozolomide or Temozolomide Followed by ATN-224 in Patients With Advanced Melanoma
Brief Title: Randomized Trial of ATN-224 and Temozolomide in Advanced Melanoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Attenuon (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ATN-224-008
Record Dates: First submitted 2006-10-02; First posted 2006-10-04 (Estimated); Last update posted 2007-12-06 (Estimated); Status verified 2007-12

CONDITIONS: Melanoma
Keywords: ATN-224; Temozolomide; Combination; Sequential; Anti-angiogenic; Copper
MeSH Terms: conditions — Melanoma | interventions — tetrathiomolybdate; Temozolomide

INTERVENTIONS:
Drug: ATN-224
Drug: Temozolomide

SUMMARY:
This is a multicenter, randomized, phase II study to evaluate the safety and efficacy of oral ATN-224 plus temozolomide in patients with advanced melanoma. Patients will be randomized (1:1) between temozolomide and ATN-224 and temozolomide followed by ATN-224. Patients assigned to the sequential treatment group will receive temozolomide until progression of disease is documented and then receive ATN-224 as a single agent until documentation of progression of disease using the last tumor assessment on temozolomide therapy as the baseline assessment.

DETAILED DESCRIPTION:
According to the National Cancer Institute PDQ database, advanced melanoma is refractory to most standard systemic therapy, and all newly diagnosed patients should be considered candidates for clinical trials. Although advanced melanoma is relatively resistant to therapy, several biologic response modifiers and cytotoxic agents have been reported to produce objective responses. Once melanoma is metastatic, treatments are palliative rather than curative. In spite of many attempts at multimodality therapy, the prognosis in this disease remains poor. Further agents are needed if progress is to be made with melanoma treatment.

ATN-224 is an orally active, small molecule that has been shown in cellular and animal models to be antiangiogenic and to have activity against melanoma cell lines. Clinical studies with a similar agent (ammonium tetrathiomolybdate) indicate that the agent can be administered continuously on a daily basis for years in some patients. ATN-224 has the potential to affect the progression of melanoma by mechanisms that include both antiangiogenic and antitumor pathways. Temozolomide, a commonly used agent for melanoma, also has a tolerable profile.

ELIGIBILITY:
Inclusion Criteria

* Patients with histologically confirmed, advanced cutaneous melanoma. Advanced melanoma is defined as locally advanced disease that is not amenable to surgery or radiation therapy and metastatic disease. Patients may have had adjuvant treatment for prior early disease as long as it was given at least 6 months before the first dose of study medication, and the treatment did not contain temozolomide or dacarbazine. Previous treatment for advanced disease is acceptable as long as the patient did not receive temozolomide or dacarbazine. There is no restriction on the number of prior regimens.
* Age ≥18 years
* Life expectancy of greater than 6 months
* Eastern Cooperative Oncology Group (ECOG) performance status ≤2 (Karnofsky ≥50%; see Appendix A)
* Patients must have adequate organ and marrow function as defined below:

  * absolute neutrophil count ≥1,500/uL
  * platelets ≥100,000/uL
  * hemoglobin ≥9 g/dL
  * total bilirubin ≤2 X institutional upper limit of normal (ULN)
  * AST(SGOT) and ALT(SGPT) ≤2 X ULN
  * creatinine clearance (measured or calculated) ≥30 mL/min

Patients are allowed to receive erythropoietin or blood transfusions before receiving their first dose of ATN-224 to bring the hemoglobin level to >9 g/dL to meet eligibility criteria.

* Use of adequate contraception. Temozolomide has the potential to cause fetal harm. The effects of ATN 224 on the developing human fetus at the recommended therapeutic dose are unknown, but antiangiogenic agents are known to be teratogenic. For these reasons women of child-bearing potential and men with partners of child-bearing potential must agree to use adequate contraception (hormonal and/or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation through the follow up visit 28 days after the last dose of ATN 224 or temozolomide.
* Willingness to forgo taking copper- or zinc-containing vitamins or supplements
* Ability to understand and the willingness to sign a written informed consent document
* Uveal (ocular) melanoma
* Brain metastasis that has not been treated and remained stable for at least 4 weeks (In other words, patients are eligible if they have no metastases or if brain metastases have been treated and remain stable for at least 4 weeks)
* Patients may not be receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to ATN-224 or omeprazole
* History of malabsorption syndromes or other gastrointestinal disorders that may affect ATN-224 or temozolomide absorption, including bowel obstruction, celiac disease, sprue, cystic fibrosis
* Ineligible to receive either temozolomide (Temodar®), omeprazole (Prilosec®), lansoprazole (Prevacid®), pantoprazole (Protonix®), or ranitidine (Zantac®)
* Inability to swallow study medication capsules
* Other serious medical or psychiatric illness preventing informed consent or with the potential to interfere with assessment of safety or efficacy of ATN-224 treatment
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Patients known to be positive for HIV or infectious hepatitis type A, B or C
* No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated Stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease-free for 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2006-09; Study Completion 2008-09 (Estimated)

PRIMARY OUTCOMES:
24-week progression-free survival of the combination of temozolomide with ATN 224 and of temozolomide alone
Evaluate the safety of ATN-224 in combination with or following temozolomide

SECONDARY OUTCOMES:
Response rate (complete and partial response), rate of stable disease for ≥24 weeks, and progression-free survival for treatment with the combination of ATN 224 and temozolomide
Response rate (complete and partial response), rate of stable disease for ≥24 weeks, and progression-free survival for treatment with temozolomide alone
Response rate (complete and partial response), rate of stable disease for ≥24 weeks, and progression-free survival for treatment with ATN 224 alone after progression of disease on temozolomide
Time to treatment failure by progression of disease or death for patients receiving ATN 224 plus temozolomide and for patients receiving temozolomide followed by ATN 224
Explore blood and tumor biomarkers with the potential to correlate with activity

CONTACTS AND LOCATIONS:
Overall Officials: Gilad Gordon, MD, Study Director
Locations (17):
- United States (17):
  - Arizona Cancer Center, Tucson, Arizona
  - Pacific Oncology and Hematology, Encinitas, California
  - Hematology - Oncology Group of Orange, Inc., Orange, California
  - UCI Chao Family Comprehensive Cancer Center, Orange, California
  - The Angeles Clinic, Santa Monica, California
  - University of Colorado Health Science Center, Denver, Colorado
  - Florida Cancer Specialists, Fort Myers, Florida
  - Hematology and Oncology Specialists, LLC, Metairie, Louisiana
  - The Harry and Jeanette Weinberg Cancer Institute at Franklin Square, Baltimore, Maryland
  - Center for Cancer and Blood Disorders, Bethesda, Maryland
  - Billings Clinic, Billings, Montana
  - Mountainside Hospital Cancer Center - The Melanoma Center, Montclair, New Jersey
  - Oncology Hematology Care, Cincinati, Ohio
  - Cancer Center of the Carolinas, Greenville, South Carolina
  - Chattanooga Oncology and Hematology Associates, Chattanooga, Tennessee
  - Tennessee Oncology, Nashville, Tennessee
  - Mary Crowley Medical Research Center, Dallas, Texas